CLINICAL TRIAL: NCT05245045
Title: Efficacy and Safety of STBF Photodynamic Therapy for Moderate and Severe Acne Vulgaris
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Dermatology Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-29
Record Dates: First submitted 2022-02-09; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Acne
Keywords: Acne; Photodynamic Therapy; Shengtaibufen; Efficacy; Safety
MeSH Terms: conditions — Acne Vulgaris | interventions — Red Light

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shengtaibufen Photodynamic Therapy(STBF-PDT) (Experimental): The Shengtaibufen photodynamic therapy group underwent narrow-band light-emitting diode (LED) irradiation (630 nm; 150 J/cm2) after applying 0.5mg/ml Shengtaibufen solution for 45min. A repeat treatment was administered once weekly for a maximum of 3 weeks.
  Interventions: Procedure: Shengtaibufen Photodynamic Therapy(STBF-PDT)
- Red light (Placebo Comparator): The Shengtaibufen photodynamic therapy group underwent narrow-band light-emitting diode (LED) irradiation (630 nm; 150 J/cm2) after applying normal saline solution for 45min. A repeat treatment was administered once weekly for a maximum of 3 weeks.
  Interventions: Procedure: Red light

INTERVENTIONS:
Procedure: Shengtaibufen Photodynamic Therapy(STBF-PDT) — Shengtaibufen Photodynamic Therapy(STBF-PDT)
  Arms: Shengtaibufen Photodynamic Therapy(STBF-PDT)
Procedure: Red light — Red light
  Arms: Red light

SUMMARY:
This study is being done to evaluate the efficacy and safety of Shengtaibufen photodynamic therapy (STBF-PDT) for treatment of moderate or severe acne vulgaris.

DETAILED DESCRIPTION:
This study is a split randomized controlled trial and being done to evaluate the efficacy and safety of Shengtaibufen photodynamic therapy (STBF-PDT) for treatment of moderate or severe acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosed with moderate to severe acne;
2. Male and female patients of age between 18-30 years old ;
3. All patients read the instructions of the subject, willing to follow the program requirements;
4. No other topical treatment received within 2 weeks prior to enrollment;
5. No systemic treatment was given within 4 weeks prior to enrollment;
6. Patients were unsuitable for surgery for various reasons,unwilling to undergo surgery, and signed informed consent when they had informed other alternatives and agreed to take pictures of the lesion.

Exclusion Criteria:

1. Those who did not complete the informed consent;
2. The lesions belongs to any of the following conditions: There is damage and inflammation, which may lead to the drug entering the open wound;
3. Patients with skin photoallergic diseases, porphyria;
4. Known to have a history of allergies to test drugs (porphyrins) and their chemically similar drugs;
5. Patients with other obvious diseases that may affect the evaluation of efficacy;
6. Scars or patients with a tendency to form scars;
7. Known to have severe immune dysfunction, or long-term use of glucocorticoids and immunosuppressants;
8. Severe heart, liver, kidney disease; with hereditary or acquired People with sexual coagulopathy
9. Those with severe neurological, psychiatric or endocrine diseases; (10)Women who are pregnant, breast-feeding or using inappropriate contraceptives; those with a history of drug abuse; those who have participated in other drug clinical trials within 4 weeks before treatment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-02-10 (Estimated); Study Completion 2023-02-10 (Estimated)

PRIMARY OUTCOMES:
The clearance rate of Moderate or Severe Acne | The clearance rate of Moderate or Severe Acne will be measured at one month after the last treatment
  The clearance rate of Moderate or Severe Acne will be measured at one month after the last treatment

SECONDARY OUTCOMES:
Adverse effect | Immediately, 1 hour, 12 hours, 24hours and 48 hours after treatment
  The pain will be assessed using Visual Analogue Scale#VAS) with a score range of 0-10. Erythema edema will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Wang, MD, Study Director — Shanghai Skin Disease Hospital
Locations (1):
- Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
study protocal
Supporting Information: CSR
Time Frame: One year after finishing this study and for permanency
Access Criteria: anyone who search pubmed